CLINICAL TRIAL: NCT02963441
Title: A Multi-center Study to Evaluate Performance of an Automated Device for the Detection of Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Digital Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IDx-DR1, version 03
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Diabetic Macular Edema; Center-involved Diabetic Macular Edema; Clinically Significant Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DME: Center-involved macular edema based on WRC of macular Optical Coherence Tomography images
  Clinically Significant macular edema based on WRC grading of widefield stereo color fundus photographs.
  Sample Size: ~45 subjects with DME
  Interventions: Device: LumineticsCore (formerly IDX-DR)

INTERVENTIONS:
Device: LumineticsCore (formerly IDX-DR) — Prospective analysis on an existing subgroup of subjects in the US pivotal study, version 01 and version 02.

SUMMARY:
Diabetes affects 30.3 million people or 9.3% of the population of the United States. Results of a study by the Eye Diseases Prevalence Research Group reveal that 40% of diabetes patients have some degree of diabetic retinopathy (DR) and that as many as 8% have severe, vision-threatening forms of DR. Early laser photocoagulation in high-risk proliferative diabetic retinopathy (PDR) has been shown to decrease the relative risk of vision loss by as much as 52%. Injections of anti-VEGF agents preserve and improve vision in people with PDR and/or diabetic macular edema. Despite effective treatment however, tens of thousands of people with diabetes are going blind each year largely because they don't undergo annual screening for retinopathy. Currently, less than 50%-60% of people with diabetes have a yearly eye exam and there may not be enough eye specialists to see the balance.

The IDx-DR System is intended for use by health care providers to automatically detect more than mild diabetic retinopathy (mtmDR) in adults (22 years of age or older) diagnosed with diabetes who have not been previously diagnosed with diabetic retinopathy. IDx-DR is indicated for use with the Topcon NW400.

DETAILED DESCRIPTION:
From January 2017 to July 2017, 900 participants were prospectively enrolled in this observational study at 10 primary care practice sites throughout the United States. The study was approved by the institutional review board for each site, and all participants provided written informed consent. The study, which was funded by IDx LLC, was designed by the authors with input from the U.S. Food and Drug Administration (FDA) on the endpoints, statistical testing, and study design. Emmes Corp, a contract research organization (CRO), provided overall project management, including data management and independent monitoring and auditing services for all sites. CCR, Inc., an Algorithm Integrity Provider (AIP), was contracted to lock the AI system, hold any intermediate and final results and images in escrow, and interdict access to these by the Sponsor, from prior to the start of the study until final data lock. Because the Sponsor was thus interdicted from access to the AI system, the AIP performed all necessary maintenance and servicing activities during the study as well as throughout closeout.

The target population was asymptomatic persons, ages of 22 and older, who had been diagnosed with diabetes and had not been previously diagnosed with DR. A diagnosis of diabetes was defined as meeting the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA); Hemoglobin A1c (HbA1c) ≥ 6.5% based on repeated assessments; Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) based on repeated assessments; Oral Glucose Tolerance Test (OGTT) with two-hour plasma glucose (2-hr PG) ≥ 200 mg/dL (11.1 mmol/L) using the equivalent of an oral 75 g anhydrous glucose dose dissolved in water; or symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L).

To help enroll a sufficient number of mtmDR participants for the evaluation of sensitivity, a stepwise enrichment strategy, as indicated in the prespecified protocol, was utilized mid-study to recruit sufficient numbers of mtmDR participants. The enrichment strategy sought higher risk participants with elevated HbA1c (>9.0%) levels or elevated Fasting Plasma Glucose; this enrichment was independently activated by the statistician while always remaining masked to the AI system outputs and the ETDRS disease levels. To account for any unintentional spectrum bias in the no/mild population, the study pre-defined a specificity outcome parameter to correct for any potential spectrum bias resulting from this enrichment strategy as co-primary.

All primary care sites in the study identified one or more inhouse operator trainees to perform the AI system protocol. After installation of the equipment by the Sponsor at the site, but before any participant was recruited, AI system operator trainees had to attest that they had not previously performed ocular imaging. Also, before start of study recruitment at each site, AI system operator trainees underwent a one-time standardized 4 h training program. They were trained how to acquire images, how to improve image quality if the AI system gave an insufficient quality output, and how to put images for analysis into the AI system. No additional training was provided to any of the AI system operators for the duration of the study. Independently, FPRC certified expert photographers were identified in geographic locations close to each site by the CRO, and documented 4W-D FPRC certification was required before any participant was imaged. The CRO independently completed site initiation visits at each site to ensure each site met all the good clinical practice requirements prior to start of enrollment.

Study protocol. All participants gave written informed consent to participate in both the AI system protocol, as well as the FPRC imaging protocol, using two different cameras:

The AI system protocol consisted of the following steps:

1. Operator takes images with a nonmydriatic retinal camera (NW400, Topcon Medical Systems, Oakland, NJ) according to a standardized imaging protocol with one disc and one fovea centered 45° image per eye;
2. Operator submits images to the AI system for automated image quality and protocol adherence evaluation;
3. If the AI system outputs insufficient quality, steps 1-2 are repeated until sufficient quality is output or 3 attempts were made. If the AI system still indicates that images are of insufficient quality, the participant's pupils are dilated with tropicamide 1.0% eyedrops, (provided by the Sponsor at each site), until the pupil diameter is at least 5mm in each eye or 30 minutes have passed, and steps 1-2 are repeated until sufficient quality is output or 3 attempts were made. If the AI system still outputs that images are of insufficient quality, the AI system output of insufficient quality is automatically provided to the CRO via secure data transfer;
4. Whenever the AI system indicates sufficient quality, the AI system disease level output (either mtmDR detected or mtmDR not detected) is automatically provided to the CRO via secure data transfer; the final AI system output provided to the CRO after this protocol was mtmDR detected, mtmDR not detected or insufficient quality

The FPRC imaging protocol was then conducted, and consisted of the following steps, all performed by an FPRC certified photographer:

1. If participant is not already dilated, dilating eye drops of tropicamide 1.0% are administered;
2. Digital widefield stereoscopic fundus photography is performed, using a camera capable of widefield photography, (Maestro, Topcon Medical Systems, Oakland, NJ) according to the FPRC 4W-D stereo protocol, by an FPRC certified photographer;
3. Anterior segment photography for media opacity assessment is performed according to the Age Related Eye Disease Study, by an FPRC certified photographer;
4. OCT of the macula is performed using a standard OCT system capable of producing a cube scan containing at least 121 B scans, (Maestro, Topcon Medical Systems, Oakland, NJ) according to the FPRC OCT protocol, by an FPRC certified photographer.

The FPRC certified photographers were masked to the AI system outputs at all times.

Reference standards. The FPRC grading protocol consisted of determination of ETDRS Severity Scale (SS) levels for fundus photographs and standardized OCT grading, as follows: the 4W-D images were read by three experienced and validated readers at the FPRC according to the well established ETDRS SS, using a majority voting paradigm. The macular OCT images were evaluated for the presence of center-involved DME by experienced readers at the FPRC according to the DRCR grading paradigm. For each participant, the ETDRS levels were mapped to mtmDR+(ETDRS level 35 or higher and /or DME present), or mtmDR- (ETDRS level 10-20 and DME absent), taking the worst of two eyes to correspond to the outputs of the AI system at the participant level.16 To measure sensitivity for the cases requiring immediate followup, called vision threatening DR, we defined vtDR + as ETDRS level 53 or higher, and/ or DME present, See Supplemental Table 2 for the mapping from ETDRS and DME levels to dichotomous mtmDR- and mtmDR +and vtDR+. Because DME can be identified both on the basis of retinal thickening on stereoscopic fundus photographs, as well as on the basis of retinal thickening on OCT, we separately analyzed both. Stereoscopic fundus based Clinically Significant DME (CSDME) was identified if there was either retinal thickening or adjacent hard exudates < 600 μm from the foveal center, or a zone of retinal thickening > 1 disc area, part of which is less than 1 disc diameter from the foveal center, according to the FPRC, in any eye. OCT based center-involved DME was identified if a participant had central subfield (a 1.0mm circle centered on the fovea) thickness that was >300 μm according to the FPRC, in any eye.20 Accordingly, we further specify the definition of mtmDR where relevant:

fundus mtmDR+ is defined as

* ETDRS level ≥ 35 (determined from fundus photographs)and/or
* CSDME (determined from fundus photographs)

and multimodal mtmDR+is defined as:

* ETDRS level ≥ 35 (determined from fundus photographs), and / or
* CSDME (determined from fundus photographs) and / or
* center-involved DME (determined from OCT).

and similarly for vtDR + . FPRC readers were masked to the AI system outputs at all times, masked to the fundus photograph reading when evaluating the OCT images, and masked to OCT readings when evaluating fundus photographs.

On September 12, 2023, Digitial Diagnostics received IRB exemption to conduct a retrospective confirmatory analysis. The pivotal study protocol was amended from version 02 to version 03 to add a prospective analysis for detecting center-involved and clinically significant DME with LumineticsCore. The level I reference standard for these forms of DME was preregistered in Version 1 of the study:

* Center-involved macular edema based on WRC of macular Optical Coherence Tomography images
* Clinically Significant macular edema based on WRC grading of widefield stereo color fundus photographs.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of diabetes mellitus, e.g.:

   1. Having met the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA)
   2. Hemoglobin A1c (HbA1c) ≥ 6.5%
   3. Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L)
   4. Oral Glucose Tolerance Test (OGTT) with two-hour plasma glucose (2-hr PG) ≥ 200 mg/dL (11.1 mmol/L), using the equivalent of an oral 75 g anhydrous glucose dose dissolved in water
   5. Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L)
2. Age 22 or older
3. Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

1. Persistent vision loss, blurred vision, or floaters.
2. Diagnosed with macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion.
3. History of laser treatment of the retina or injections into either eye, or any history of retinal surgery.
4. Currently participating in another investigational eye study and actively receiving investigational product for DR or DME.
5. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation).
6. Participant is contraindicated for imaging by fundus imaging systems used in the study:

   * Participant is hypersensitive to light
   * Participant recently underwent photodynamic therapy (PDT)
   * Participant is taking medication that causes photosensitivity

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic - sampling method: non-probability sequential, invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abramoff MD, Lavin PT, Birch M, Shah N, Folk JC. Pivotal trial of an autonomous AI-based diagnostic system for detection of diabetic retinopathy in primary care offices. NPJ Digit Med. 2018 Aug 28;1:39. doi: 10.1038/s41746-018-0040-6. eCollection 2018. PMID 31304320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2017 to July 2017, 900 participants were prospectively enrolled in this observational study at 10 primary care practice sites throughout the United States.
Groups:
- Intent to Screen Population: Prospective study participants
Period: Overall Study
Arm/Group | Intent to Screen Population
Started | 900
Completed | 819
Not Completed | 81
Not completed — Protocol violation or withdrawn | 8
Not completed — Ungradeable by FPRC or IDx | 40
Not completed — IDx-DR insufficient quality | 33

BASELINE CHARACTERISTICS:
Population: Number of analyzable study participants
Groups:
- Effective Analysis Population: All subjects with a reading center reference standard and AI output (population that is available for statistical analysis).
Arm/Group | Effective Analysis Population
Number analyzed (Participants) | 819
Age, Categorical [Count of Participants; unit: Participants]
  Age (years): <=18 years | 0
  Age (years): Between 18 and 65 years | 566
  Age (years): >=65 years | 253
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 389
  Female | 430
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 134
  Not Hispanic or Latino | 680
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 231
  White | 523
  More than one race | 10
  Unknown or Not Reported | 40
Region of Enrollment [Number; unit: participants]
  United States | 819

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity Corrected for Enrichment
Description: Sensitivity corrected for enrichment using logistic regression
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Groups:
- Analyzable Study Population: Participants that had reading center grading and AI disease outputs that were available for statistical analysis.
Arm/Group | Analyzable Study Population
Number analyzed (Participants) | 819
percentage of true positives | 87.2 [81.8 to 91.2]

2. Primary Outcome: Specificity Corrected for Enrichment
Description: Specificity corrected for enrichment using logistic regression
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Analyzable Study Population
Number analyzed (Participants) | 819
percentage of true negatives | 90.7 [88.3 to 92.7]

3. Primary Outcome: Observed Sensitivity
Description: The sensitivity observed without adjustment by logistic regression
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Analyzable Study Population
Number analyzed (Participants) | 819
percentage of true positives | 87.4 [81.9 to 92.9]

4. Primary Outcome: Observed Specificity
Description: The specificity observed without adjustment by logistic regression
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Analyzable Study Population
Number analyzed (Participants) | 819
percentage of true negatives | 89.5 [86.9 to 93.1]

5. Primary Outcome: Sufficient vs. Insufficient Image Quality Output From IDx-DR
Description: Image-ability, defined as the percentage of participants with a completed reading center grading and a disease level output from the investigational device (IDx-DR)
Time Frame: Day 1
Population: Image-ability, defined as the percentage of participants with a completed FPRC grading and a disease level IDx-DR output
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Analyzable Study Population: Participants with the reading center results needed for study analysis.
Arm/Group | Analyzable Study Population
Number analyzed (Participants) | 852
percentage of participants | 96.1 [94.0 to 96.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 to 30 days after last study contact.
Groups:
- Enrolled Population: All study subjects enrolled into the clinical study.
Arm/Group | Enrolled Population
All-Cause Mortality (participants affected / at risk) | 0/900
Serious Adverse Events (participants affected / at risk) | 0/900
Other Adverse Events (participants affected / at risk) | 5/900
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Population (N=900)
Panic attack (Psychiatric disorders) | 1 (1) — symptoms occurred after eye drops instilled
Hypoglycemic Episode (Metabolism and nutrition disorders) | 1 (1)
Eye edema (Eye disorders) | 1 (1) — Bilateral swelling in eyes post dilation
Hypotension (Vascular disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) — burning sensation
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study, Institution will be free to publish the methods, data and results of the Study

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02963441/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02963441/SAP_001.pdf